CLINICAL TRIAL: NCT01813825
Title: A Single Site Prospective, Non-randomized Study of Partial Breast Intracavitary Brachytherapy Devices to Evaluate Local Tumor Control, Cosmetic Outcome and Toxicities.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Vincent's Medical Center (Unknown)
Responsible Party: Principal Investigator, Deborah Fang, MD, Radiation Oncology, St. Vincent's Medical Center
Organization: St Vincent's Hospital (Other)
Other Study IDs: SVMC 104
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: This Study Has Been Designed to Compile Information on the Efficacy of the Partial Breast Intracavitary Brachytherapy in the Post Market Setting.
Keywords: Mammosite
MeSH Terms: interventions — Registries

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Female >=45 years, negative margins, DCIS
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry

SUMMARY:
A registry is an observation database. Participation in this registry does not require any additional or different procedures or drugs other than those you would normally receive for breast cancer. Registry databases are used to identify trends in medical care that help the medical community identify optimal care for different diseases.

The data will be compiled on the safety and performance of the Partial Breast Brachytherapy Applicator based on the information collected about the treatment and follow up visits.

DETAILED DESCRIPTION:
PURPOSE OF STUDY

The patient understand that she has cancer of the breast. The patient understand that is offered the opportunity to participate in a registry study to collect data on the FDA approved device,Partial Breast Brachytherapy Applicator. Partial Breast Brachytherapy is a treatment method that works by delivering radiation from inside the breast directly to the tissue where cancer is most likely to recur. The Partial Breast Brachytherapy Applicator is a device that has tiny catheters or wires that fit inside the lumpectomy cavity (the space left after the tumor is removed). Radioactive sources (seed) are placed within the device by a computer controlled machine. This radioactive source will deliver the radiation therapy to the breast

A registry is an observation database. Participation in this registry does not require any additional or different procedures or drugs other than those you would normally receive for breast cancer. Registry databases are used to identify trends in medical care that help the medical community identify optimal care for different diseases.

PROCEDURES

If the patient agree to take part in this registry, data will be compiled on the safety and performance of the Partial Breast Brachytherapy Applicator based on the information collected about the treatment and follow up visits.

POTENTIAL RISKS AND DISCOMFORTS

There is no medical risk to the patient if she takes part in this registry, as she will continue to receive the same medical care as provided by her medical team.

POTENTIAL BENEFITS:

It is not possible to state that the patient will benefit from this study. The information obtained from study may be used scientifically and may possibly be helpful to others.

ALTERNATIVES TO TREATMENT

The patient participation is voluntary and she may choose not to participate in this study or she may stop at any time. The patient choice will not affect doctors from providing care. The patient will not lose any benefits if she choose not to participate or if you withdraw from this study. She is free to seek care from a doctor of her choice at any time.

ELIGIBILITY:
Inclusion Criteria:

* Be 45 years of age or older
* Be a Tis, T1, N0 M0 - American Joint Committee Classification
* Have negative surgical margins (NSABP definition) after final surgery
* Should have adequate skin spacing between balloon surface and surface of the skin (>=7mm)
* DCIS

Exclusion Criteria:

* Be pregnant or breast-feeding.(If appropriate, patient must use birth control during the study)
* Have collagen-vascular disease
* Have extensive intraductal component (Harvard Definition,>25% DCIS)
* Have infiltrating lobular histology

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females, with Breast Cancer Tis, T1,N0,M0. Negative Surgival Margens
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2004-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
A Single Site Prospective, Non Randomized Study of Partial Breast Intracavitary Brachytherapy Devices To Evaluate Local Tumor Control, Cosmetic Outcome and Toxicities | 1-4 weeks
  The efficacy of the treatment will be measured by using the overall survival. The following endpoints will also be reported and analyzed:Disease Free Survival, Cause Specific Survival, Ipsilateral Breast Failure, Contralateral Breast Failure.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Fang, MD, Principal Investigator — St. Vincent's Medical Center
Locations (1):
- St. Vincent's Medical Center, Bridgeport, Connecticut, United States